CLINICAL TRIAL: NCT05656690
Title: Study and Analysis of Biomechanical Parameters of Human Movement Based on Disability Indicators in Older Adults Based on a Multifactorial Analysis: a Prospective Cohort Study
Brief Title: Prospective Study and Analysis of Biomechanical Parameters of Human Movement Based on Disability Indicators in Older Adults
Acronym: MOBA-P
Status: Completed | Type: Observational
Sponsor: Polytechnic Institute of Porto (Other)
Collaborators: Center for Rehabilitation Research - Polytechnic Institute of Porto (IPP) (Unknown); Universidade do Porto (Other); School of Allied Health Sciences of Porto (ESTSP) - Polytechnic Institute of Porto (IPP) (Other)
Responsible Party: Principal Investigator, Juliana dos Santos Moreira, PhD grant student, Polytechnic Institute of Porto
Other Study IDs: CE0077C; 2020.05356.BD (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia, Portugal, NORTE 2020, FSE EU); UIDB/05210/2020 (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia (FCT), Portugal and the European Union (EU))
Record Dates: First submitted 2022-11-18; First posted 2022-12-19 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy older Adults: Healthy older Adults: older adults without disability indicators
  Interventions: Other: Exposure to disability
- Disability Older Adults: Disability Older Adults: older adults with disability indicators
  Interventions: Other: Exposure to disability

INTERVENTIONS:
Other: Exposure to disability — Disability status assessed by functional measures

SUMMARY:
Mobility loss in older people is caused by a variety of aging impairments in various body systems.The disability, which includes physical impairments and resulting activity limitations or participation restrictions, can arise acutely from a catastrophic illness or, more commonly, from subacute functional decline without a clear triggering event. Lower physical functioning was associated with higher healthcare utilization and expenditures, leading to a large burden on government-funded healthcare services. Early identification of mobility changes and intervening in them would likely be the most effective strategy to reduce the burden of disability in the population. Overall, there is a need to develop strategies to reduce disability among older adults in which kinetic and kinematic characteristics are used to predict disability status.

Accordingly, the purpose of this prospective cohort is to identify biomechanical parameters, from the gait, sit-to-stand, timed up and go, stair ascend and descend, and quiet standing functional tasks, as predictors of changes in health and disability status in older adults.

This research was funded by Fundação para a Ciência e Tecnologia (FCT), NORTE 2020, and European Social Fund of European Union, grant number 2020.05356.BD and through R&D Units funding (UIDB/05210/2020), Fundação para a Ciência e Tecnologia (FCT), Portugal and the European Union.

ELIGIBILITY:
Inclusion Criteria:

* older adults, 60 years or over;
* community-dwelling;
* able to perform the tasks (gait, sit-to-stand, climb and descend stairs) independently;

Exclusion Criteria:

* older adults who are institutionalized;
* older adults who have established diagnosis of malignancy or terminal diseases with an anticipated survival of less than 1 year;
* older adults who have stroke history, cerebral hemorrhage, head trauma, or Parkinson's disease;
* older adults who have cognitive impairment, specifically Mini Mental StateExamination (Portuguese version) score of 22 for 0 to 2 years of literacy, 24 for 3 to6 years of literacy and 27 for more than 6 years of literacy (Morgado et al., 2009);
* older adults who have rheumatic pathologies that interfere with the tasks performance;
* older adults who have diabetic foot, lower limb fracture less than 6 weeks, or other related conditions;
* older adults who have unstable cardiovascular disease, liver or renal function failure;
* older adults who have a body mass index greater than or equal to 30 kg/m2;
* older adults who vestibular and/or audition or vision impairments non corrected that influence the performance of tasks;
* older adults who presence of symptoms at the time of evaluation that influences the participant performance of tasks.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Portuguese community-dwelling older adults
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Waveforms from full-body joint angles | Assessed once at study entry.
  Waveforms from full-body joint angles measured in degrees (°)
Waveform from full-body angular joint velocities | Assessed once at study entry
  Waveform from angular joint velocities measured in degrees per second (°/s)
Waveform from lower limb joint moments | Assessed once at study entry
  Waveform from lower limb joint moments measured in Newton-meter (kgm²/s²)
Waveform from total body energy | Assessed once at study entry
  Waveform from total body energy measured in joules (J)
Waveform from full-body separate segment energy | Assessed once at study entry
  Waveform from body segment energy un joules (J)
Waveform from lower body joint forces | Assessed once at study entry
  Waveform from lower body joint forces measured in Newton (N)
Waveform from lower body joint power | Assessed once at study entry
  Waveform from lower body joint power measured in Watts
Waveform from centre of mass displacement | Assessed once at study entry
  Waveform from centre of mass displacement in m/s
Waveform from centre of pressure displacement | Assessed once at study entry
  Waveform from centre of pressure displacement in m/s
International Physical Activity Questionnaire | Assessed at study entry and evaluated every three months until the end of 1 year
  IPAQ is questionnaire to assess self-reported physical activity
Mini-Mental State Examination (MMSE) | Assessed at study entry and evaluated every three months until the end of 1 year
  MMSE provides a brief screening test that quantitatively assesses the severity of cognitive impairment and documents cognitive changes occurring over time
Barthel Index | Assessed at study entry and evaluated every three months until the end of 1 year
  The Barthel Index is an instrument that assesses the individual's level of independence for ten activities of daily living
Lawton and Brody Instrumental Activities of Daily Living Scale | Assessed at study entry and evaluated every three months until the end of 1 year
  Lawton and Brody Instrumental Activities of Daily Living Scale assess the instrumental ADLs necessary for living in the community
Number of health conditions | Assessed at study entry and evaluated every three months until the end of 1 year
  Total number and description of health conditions
Number of falls | Assessed at study entry and evaluated every three months until the end of 1 year
  Total number and description of ocurrences of falls

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Rehabilitation Research, School of Health, Polytechnic of Porto, Portugal, Porto, Portugal